CLINICAL TRIAL: NCT04894422
Title: Effect of Face Masks on the Microbial Communities of the Skin and Upper Airways and the Optimalisation of Microbiome Analysis
Brief Title: Microbiome Analysis of Skin and Airway Samples and Effect of Face Masks
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Sarah Lebeer, Principal Investigator, University Hospital, Antwerp
Other Study IDs: B3002021000072
Record Dates: First submitted 2021-05-11; First posted 2021-05-20 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Healthy
Keywords: skin microbiome; 16S amplicon sequencing; face masks; upper airway microbiome; shotgun sequencing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Isolation of microbial DNA and/or RNA out of skin and upper airway swabs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- No face mask: Volunteers who did not wear a face mask
  Interventions: Other: Observational intervention
- Cotton face mask: Voluntarily wearing a cotton face mask for 4 hours, following the government's guidelines during the COVID-19 pandemic.
  Interventions: Other: Observational intervention
- Surgical face mask: Voluntarily wearing a surgical face mask for 4 hours, following the government's guidelines during the COVID-19 pandemic.
  Interventions: Other: Observational intervention

INTERVENTIONS:
Other: Observational intervention — Voluntarily (not) wearing a face mask (cotton or surgical) for 4 hours, following the government's guidelines during the COVID-19 pandemic.

SUMMARY:
The goal of this study is to optimize two methods for microbiome analysis of skin and upper airway samples (16S amplicon sequencing and Shotgun sequencing). In addition, the researchers will investigate whether there is an effect of wearing a face mask on the microbial communities of the skin and upper airways. The volunteers will self-collect swabs of the skin and upper airways (nose and/or throat). Bacterial DNA and/or total RNA will be isolated and the microbial communities will be investigated with 16S amplicon sequencing and shotgun metagenomic sequencing.

ELIGIBILITY:
Inclusion Criteria:

* Adult age 18 at the start of the study

Exclusion Criteria:

* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy, adult volunteers
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-03-15 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2023-03-15 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in microbiome composition of the skin and upper airways after wearing a face mask | Start, 4 hours
  16S rRNA sequencing
Optimalization of microbiome analysis of skin and upper airway samples | Start
  16S rRNA sequencing, shotgun metagenomic sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Lebeer, Prof., Principal Investigator — Universiteit Antwerpen
Locations (1):
- University of Antwerp and University Hospital Antwerp, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No